CLINICAL TRIAL: NCT00706173
Title: A Randomized Double-blind Placebo-controlled Cross-over Trial of Hydrocortisone for Post-traumatic Stress Disorder
Brief Title: Trial of Hydrocortisone for Post-Traumatic Stress Disorder (PTSD)
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to recruit eligible subjects for the trial.
Sponsor: University of California, San Diego (Other)
Responsible Party: Murray B. Stein, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 071982
Record Dates: First submitted 2008-06-25; First posted 2008-06-27 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2011-08

CONDITIONS: Post-traumatic Stress Disorder
Keywords: Post-traumatic stress disorder; PTSD; Cortisol; hydrocortisone; pharmacological treatment
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hydrocortisone (Experimental)
  Interventions: Drug: Hydrocortisone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydrocortisone — Hydrocortisone 10-20 mg PO daily for 4 weeks.
  Other Names: cortisol
  Arms: Hydrocortisone
Drug: Placebo — Placebo "10-20 mg" PO daily for 4 weeks.
  Arms: Placebo

SUMMARY:
Developing novel and effective pharmacologic interventions for this post-traumatic stress disorder is important. The investigators propose to replicate findings of an earlier published pilot study using low dose hydrocortisone as a treatment for PTSD. In order to do so in a more meaningful way, the investigators will conduct a larger but similar randomized double-blind placebo-controlled, cross-over design treatment study examining the use of low dose hydrocortisone (or placebo) for 4 weeks in combat veterans suffering from PTSD.

The investigators hypothesize that, as described by Aerni et al. (2004), administration of daily hydrocortisone will lead to a reduction in PTSD symptom severity, but particularly for re-experiencing types (e.g., flashbacks, nightmares)of symptoms. The investigators also hope to examine potential predictors and moderators of treatment response based on subjects' clinical characteristics, as well as serum cortisol and ACTH levels.

ELIGIBILITY:
Inclusion Criteria:

* Male military veterans
* Between the ages of 18-65 years old
* Generally good medical health with no clinically significant abnormalities on physical examination, electrocardiogram, or laboratory findings
* Ability to provide informed consent and comply with requirements of study protocol
* No specific contraindications to hydrocortisone
* Clinically predominant DSM-IV diagnosis of PTSD
* Score of ≥ 40 on Clinician Administered PTSD Scale [CAPS]

Exclusion Criteria:

* History of moderate to severe traumatic brain injury, seizure or organic mental illness
* Lifetime history of schizophrenia, bipolar disorder, other psychotic disorder, or depression with a score of ≥ 16 on the 17-item Hamilton Depression Rating Scale (Hamilton, 1960), active suicidal ideation
* Unstable medical illness
* Subjects undergoing any formal psychotherapy within 3 months of enrollment
* Subjects that meet criteria for substance dependence during the last 6 months
* History of adverse reaction to corticosteroids.
* Concurrent use of other psychotropic medication (e.g. benzodiazepines, antipsychotics)

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-08; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale (CAPS) | Week 0,2,4,6,8,10
Clinical Global Impressions - Improvement (CGI-I) | Week 0,2,4,6,8,10

SECONDARY OUTCOMES:
Sheehan Disability Inventory (SDI) | Week 0,4,6,10
Brief Symptom Inventory - 18 item (BSI-18) | Week 0,2,4,6,8,10

CONTACTS AND LOCATIONS:
Overall Officials: Murray B Stein, MD, MPH, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

REFERENCES:
- [Background] Aerni A, Traber R, Hock C, Roozendaal B, Schelling G, Papassotiropoulos A, Nitsch RM, Schnyder U, de Quervain DJ. Low-dose cortisol for symptoms of posttraumatic stress disorder. Am J Psychiatry. 2004 Aug;161(8):1488-90. doi: 10.1176/appi.ajp.161.8.1488. PMID 15285979
- [Background] Schelling G, Briegel J, Roozendaal B, Stoll C, Rothenhausler HB, Kapfhammer HP. The effect of stress doses of hydrocortisone during septic shock on posttraumatic stress disorder in survivors. Biol Psychiatry. 2001 Dec 15;50(12):978-85. doi: 10.1016/s0006-3223(01)01270-7. PMID 11750894
- [Background] Schelling G, Kilger E, Roozendaal B, de Quervain DJ, Briegel J, Dagge A, Rothenhausler HB, Krauseneck T, Nollert G, Kapfhammer HP. Stress doses of hydrocortisone, traumatic memories, and symptoms of posttraumatic stress disorder in patients after cardiac surgery: a randomized study. Biol Psychiatry. 2004 Mar 15;55(6):627-33. doi: 10.1016/j.biopsych.2003.09.014. PMID 15013832
- [Background] Olff M, Guzelcan Y, de Vries GJ, Assies J, Gersons BP. HPA- and HPT-axis alterations in chronic posttraumatic stress disorder. Psychoneuroendocrinology. 2006 Nov;31(10):1220-30. doi: 10.1016/j.psyneuen.2006.09.003. Epub 2006 Nov 1. PMID 17081699
- See also: UCSD Anxiety Disorders Research Program — http://www.veryshy.org